CLINICAL TRIAL: NCT02507206
Title: A D1 Agonist For Working Memory Enhancement In The Schizophrenia Spectrum
Brief Title: A D1 Agonist For Working Memory
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antonia New (Other)
Collaborators: New York State Psychiatric Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Antonia New, Professor of Psychiatry and Director of Medical Student Education, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 11-1279; 5R01MH097799-02 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Schizotypal Personality Disorder; SPD
Keywords: schizotypal personality disorder; cognitive impairment; working memory; Dopamine Agonists; Cognition Disorders; Personality Disorders; Delirium; Dementia; Amnestic; Cognitive Disorders; Mental Disorders; Dihydrexidine; Dopamine A
MeSH Terms: conditions — Schizotypal Personality Disorder; Cognitive Dysfunction; Cognition Disorders; Personality Disorders; Delirium; Dementia; Mental Disorders | interventions — dihydrexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DAR 0-100A then Placebo (Experimental): 15 mg is dissolved in 150 cc NS administered over 30 minutes x 3 consecutive days. Subjects will return a minimum of two weeks later for Visit 5 to receive drug (if randomized initially to placebo) or placebo (if randomized to drug).
  Interventions: Drug: DAR 0-100A; Drug: Placebo
- Placebo then DAR 0-100A (Placebo Comparator): 15 mg dissolved in 150 cc NS saline is administered over 30 minutes x 3 consecutive days. Subjects will return a minimum of two weeks later for Visit 5 to receive drug (if randomized initially to placebo) or placebo (if randomized to drug).
  Interventions: Drug: DAR 0-100A; Drug: Placebo
- Healthy Control (No Intervention): patients without diagnosis of SPD

INTERVENTIONS:
Drug: DAR 0-100A — 15 mg DAR 0100A is dissolved in 150 cc NS administered over 30 minutes intravenously.
  Other Names: DHX; dihydrexidine
  Arms: DAR 0-100A then Placebo; Placebo then DAR 0-100A
Drug: Placebo — 15 mg DAR placebo is dissolved in 150 cc NS administered over 30 minutes intravenously.
  Arms: DAR 0-100A then Placebo; Placebo then DAR 0-100A

SUMMARY:
The purpose of the study is to examine the effects of the administration of a drug called DAR-0100A on attention and memory in persons with schizotypal personality disorder (SPD). DAR-0100A has not been FDA approved, however in recent studies has been used to treat cognitive deficits, meaning problems in the way you organize your thinking, in people diagnosed with schizophrenia.

Many people who carry a diagnosis of schizotypal personality disorder have trouble with attention and memory. Increasing the presence of a brain chemical called dopamine has been found to help people with schizophrenia with their attention and memory problems. This study will investigate whether the same is true for people with schizotypal personality disorder by using DAR-0100A, a drug that has been shown to help with the cognitive deficits of people with Parkinson's disease by increasing dopamine effects. Information collected in this experiment may lead to a better understanding of the brain mechanisms involved in schizotypal personality disorder and improve treatments for the psychological problems associated with this condition.

DETAILED DESCRIPTION:
Primary Aims:

1. To perform a 5-year study in which three consecutive days of DAR-0100A at a dose of 15 mg or placebo are administered intravenously over 30 minutes to 60 patients with SPD (12/yr) in a between-groups, randomized, double-blind design. Cognitive testing will be performed at baseline (Visit 1) and on the third day of drug/placebo administration (Visit 4). Subjects will return a minimum of two weeks later for Visit 5 to receive drug (if randomized initially to placebo) or placebo (if randomized to drug) in a double blind fashion in an identical protocol. This allows all patients to receive drug for Secondary Aim 1 while maintaining the blind. Baseline (Visit 1) and repeat cognitive testing (Visit 4) is also administered to 60 healthy controls per year (12/yr). The cognitive tests of working memory serving as primary outcome measures will include the modified AX-CPT (accuracy scores for AX, AY and BX and ANOVA), the N-back (delta difference 0-back-2-back), and the Paced Auditory Serial Addition Task (PASAT) (% correct and ANOVA). Other tests included are tests of working and verbal memory, executive function, and verbal learning for secondary outcome measures as well as comparison tests not hypothesized to change with drug.
2. To compare changes on the primary outcome measures from baseline to Visit 4 testing between drug and placebo administration in SPD subjects.
3. To compare primary outcome variables from baseline to Visit 4 between patients groups and healthy controls.
4. To obtain plasma DAR-0100A concentrations on Visit 4 to evaluate plasma concentrations in relation to cognitive changes as a potential covariate.

Secondary Aims:

1. To evaluate the change between baseline and Visit 4 cognitive testing in all SPD patients receiving drug in the first or second phase.
2. To evaluate secondary outcome and comparison variables between SPD patients on placebo and drug.

Primary Hypotheses:

1. Baseline primary outcome measures will be impaired in SPD subjects compared to controls. 2. SPD subjects on DAR-0100A will show improvement on primary measures greater than healthy controls and SPD patients randomized to placebo between baseline and Visit 4.

3. SPD patients will show significant improvements on primary outcome variables on drug compared to placebo but not on comparis-on perceptual (JLOT) and processing speed/attentional tasks (Trails A).

ELIGIBILITY:
Inclusion Criteria:

* Currently meeting DSM-IV-TR criteria for Schizotypal
* Personality Disorder
* Males and Females 18 ≤ age ≤ 65
* Medically and neurologically healthy
* Willing and having capacity to provide informed consent

Exclusion Criteria:

* Currently bipolar I disorder, schizophrenia or current psychosis
* Clinically significant cardiovascular or neurological conditions, uncontrolled hypertension, clinically significant EKG abnormalities, or serious general medical illness
* Clinical evidence of dehydration or significant hypotension
* Currently meeting DSM-IV-TR criteria for Major Depressive Disorder
* Current substance abuse or past dependence within the last six months (other than nicotine)
* Currently taking psychotropic medications
* Currently pregnant or lactating
* Non-English speaking
* Socio-economically disadvantaged people will be included in our research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
The Modified AX-CPT (d') | Baseline performance
  A cognitive test of working memory

SECONDARY OUTCOMES:
The Modified AX-CPT (d') | Day one
  A cognitive test of working memory
The Modified AX-CPT (d') | Day three
  A cognitive test of working memory
The Modified AX-CPT (d') | One month
  A cognitive test of working memory

OTHER OUTCOMES:
the N-Back | Baseline
  A cognitive tests of working memory - the N-Back (% correct at the 2-back condition)
the N-Back | Day one
  A cognitive tests of working memory - the N-Back (% correct at the 2-back condition)
the N-Back | Day three
  A cognitive tests of working memory - the N-Back (% correct at the 2-back condition)
the N-Back | One month
  A cognitive tests of working memory - the N-Back (% correct at the 2-back condition)
the DOT Task | Baseline
  A cognitive tests of working memory - the DOT Task (distance error at 30 second delay--no delay)
the DOT Task | Day one
  A cognitive tests of working memory - the DOT Task (distance error at 30 second delay--no delay)
the DOT Task | Day three
  A cognitive tests of working memory - the DOT Task (distance error at 30 second delay--no delay)
the DOT Task | One month
  A cognitive tests of working memory - the DOT Task (distance error at 30 second delay--no delay)
the Paced Auditory Serial Addition Task (PASAT) | Baseline
  A cognitive tests of working memory - the Paced Auditory Serial Addition Task
the Paced Auditory Serial Addition Task (PASAT) | Day one
  A cognitive tests of working memory - the Paced Auditory Serial Addition Task
the Paced Auditory Serial Addition Task (PASAT) | Day three
  A cognitive tests of working memory - the Paced Auditory Serial Addition Task
the Paced Auditory Serial Addition Task (PASAT) | One month
  A cognitive tests of working memory - the Paced Auditory Serial Addition Task

CONTACTS AND LOCATIONS:
Overall Officials: Antonia S. New, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Arnsten AF, Cai JX, Murphy BL, Goldman-Rakic PS. Dopamine D1 receptor mechanisms in the cognitive performance of young adult and aged monkeys. Psychopharmacology (Berl). 1994 Oct;116(2):143-51. doi: 10.1007/BF02245056. PMID 7862943
- [Background] Abi-Dargham A. Probing cortical dopamine function in schizophrenia: what can D1 receptors tell us? World Psychiatry. 2003 Oct;2(3):166-71. PMID 16946930
- [Background] Castner SA, Williams GV, Goldman-Rakic PS. Reversal of antipsychotic-induced working memory deficits by short-term dopamine D1 receptor stimulation. Science. 2000 Mar 17;287(5460):2020-2. doi: 10.1126/science.287.5460.2020. PMID 10720329
- [Background] Fici GJ, Wu H, VonVoigtlander PF, Sethy VH. D1 dopamine receptor activity of anti-parkinsonian drugs. Life Sci. 1997;60(18):1597-603. doi: 10.1016/s0024-3205(97)00126-4. PMID 9126882
- [Background] Kirrane RM, Mitropoulou V, Nunn M, New AS, Harvey PD, Schopick F, Silverman J, Siever LJ. Effects of amphetamine on visuospatial working memory performance in schizophrenia spectrum personality disorder. Neuropsychopharmacology. 2000 Jan;22(1):14-8. doi: 10.1016/S0893-133X(99)00075-5. PMID 10633486
- [Background] Koenigsberg HW, Reynolds D, Goodman M, New AS, Mitropoulou V, Trestman RL, Silverman J, Siever LJ. Risperidone in the treatment of schizotypal personality disorder. J Clin Psychiatry. 2003 Jun;64(6):628-34. doi: 10.4088/jcp.v64n0602. PMID 12823075